CLINICAL TRIAL: NCT06376331
Title: Washed Microbiota Transplantation for Attention-deficit/Hyperactivity Disorder and Its Comorbidities
Brief Title: Washed Microbiota Transplantation for Attention-deficit/Hyperactivity Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADHD20240403
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: attention-deficit/hyperactivity disorder; washed microbiota transplantation; fecal microbiota transplantation; sleep disturbance; gut-brain axis
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Washed microbiota transplantation (Experimental): WMT
  Interventions: Drug: washed microbiota transplantation

INTERVENTIONS:
Drug: washed microbiota transplantation — The prepared microbiota suspension was infused into the participates' lower gut.
  Other Names: fecal microbiota transplantation

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a common neurodevelopmental disorder characterized by inattention and hyperactivity-impulsivity. ADHD is often accompanied by oppositional defiant disorder and sleep disturbance, and can increase the risk of other psychiatric disorders, functional impairment in academic and occupational performance. Recently, gut microbiota has been implicated in the ADHD via gut-brain axis. In this study, investigators aimed to evaluate the efficacy of WMT for core ADHD symptoms and its comorbidities using specialized questionnaires for ADHD and investigate the underlying mechanism.

DETAILED DESCRIPTION:
Gut microbiota dysbiosis has been reported to play a critical role in the initiation and progression of neurodevelopmental disorders like ADHD via the gut-brain axis. Therapies targeting gut microbiota including including probiotics, prebiotics and fecal microbiota transplantation (FMT) might provide new insight into the management of ADHD. FMT has been reported to be a highly effective therapy to restore the gut microbiota dysbiosis by transferring gut microbiota from healthy donors to patients. The newly improved methodology of FMT based on the automatic washing process and the related delivering consideration was named as washed microbiota transplantation (WMT) by the FMT-standardization study group. FMT has shown treatment potential in several gut-brain axis-related disorders, such as amyotrophic lateral sclerosis and Parkinson's disease, promoting us to investigate its treatment potential for ADHD and its comorbidities. To date, only one case report showed a 22-year-old woman undergoing FMT primarily to treat recurrent Clostridioides difficile infection achieved ADHD symptoms alleviation. However, the efficacy of WMT for ADHD and the underlying mechanisms remain largely unexplored. In this study, investigators aimed to evaluate the efficacy of WMT for core ADHD symptoms and its comorbidities using specialized questionnaires for ADHD and investigate the underlying mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Children with an established diagnosis of ADHD according to Diagnostic And Statistical Manual Of Mental Disorders Fifth Edition;
2. Aged 3-17;
3. Received stable treatments for ≥1 month preceding WMT;
4. Did not take medications affecting gut microbiota such as antibiotics and probiotics three months before WMT.

Exclusion Criteria:

1. Unable to understand the questionnaires or provide informed consent by the guardian;
2. Diagnosed with a single-gene disorder, psychosis, central nervous system diseases, gastrointestinal diseases including ulcerative colitis, Crohn's disease, celiac disease, or eosinophilic esophagitis;
3. Had severe comorbidities including cardiopulmonary failure, severe liver, and kidney diseases and cancer;
4. Accompanied with other life-threatening disorders required emergency treatment;
5. Unable to tolerate colonoscopy or anesthesia

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions-Improvement (CGI-I) | 1 month, 3 months post transplantation
  The Clinical Global Impressions-Improvement (CGI-I) evaluated by experienced clinician was used to assess the symptom changes relative to baseline, rated on a 7-point scale from 1 (very much improved) to 7 (very much worse). CGI-I = 1 or 2 was considered a clinical response.

SECONDARY OUTCOMES:
change of the Sleep Disturbance Scale for Children (SDSC). | baseline, 1 month, 3 months post transplantation
  The SDSC is 26-item test measuring sleep problems and each item receives a value from 1 to 5, with higher scores indicating more severe sleep disorders.
change of the Gastrointestinal Symptom Rating Scale (GSRS) . | baseline, 1 month, 3 months post transplantation
  It is based on 15 questions which are scored into 5 domains: abdominal pain, reﬂux, indigestion, diarrhea, and constipation. Each item weights from 1 to 7, with higher scores reflecting more severe symptoms.
the difference of the gut microbe composition between children with ADHD and healthy children by sequencing faecal metagenome. | baseline, 1 month, 3 months post transplantation
  The composition of the gut microbiota is evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism between the two at the phylum, genus and species levels of the intestinal flora and control children, and to develop a model for predicting the structure of the flora.
intestinal barrier | baseline, 1 month, 3 months post transplantation
  plasma DAO, D-lactic acid and bacterial endotoxin levels
change of Swanson, Nolan and Pelham-IV (SNAP-IV). | baseline, 1 month, 3 months post transplantation
  It is an 26-item questionnaire that measured three of the ADHD symptoms, inattention, hyperactivity and oppositional defiant disorder. The 26-item checklist is scored on a 4-point Likert scale ranging between Not At All (0) and Very Much (3).
Conners' Parent Rating Scale-Revised | baseline, 1 month, 3 months post transplantation
  ADHD symptoms were also assessed by the Conners' Parent Rating Scale-Revised (CPRS-R). The CPRS-R was composed of 10 items derived from the Revised Conners Parent Rating Scale. It used a 4-point Likert scale (range: 0-30), with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - SIR RUN RUN hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faraone SV, Bellgrove MA, Brikell I, Cortese S, Hartman CA, Hollis C, Newcorn JH, Philipsen A, Polanczyk GV, Rubia K, Sibley MH, Buitelaar JK. Attention-deficit/hyperactivity disorder. Nat Rev Dis Primers. 2024 Feb 22;10(1):11. doi: 10.1038/s41572-024-00495-0. PMID 38388701
- [Background] Bansal PS, Goh PK, Southward MW, Sizemore YJ, Martel MM. Impulsivity as key bridge symptoms in cross-sectional and longitudinal networks of ADHD and ODD. J Child Psychol Psychiatry. 2024 Jan;65(1):52-63. doi: 10.1111/jcpp.13863. Epub 2023 Jul 20. PMID 37474723
- [Background] Liang X, Qiu H, Li SX. Objectively measured sleep continuity in children and adolescents with ADHD: A systematic review and meta-analysis. Psychiatry Res. 2023 Oct;328:115447. doi: 10.1016/j.psychres.2023.115447. Epub 2023 Aug 28. PMID 37657199
- [Background] Hartman CA, Larsson H, Vos M, Bellato A, Libutzki B, Solberg BS, Chen Q, Du Rietz E, Mostert JC, Kittel-Schneider S, Cormand B, Ribases M, Klungsoyr K, Haavik J, Dalsgaard S, Cortese S, Faraone SV, Reif A. Anxiety, mood, and substance use disorders in adult men and women with and without attention-deficit/hyperactivity disorder: A substantive and methodological overview. Neurosci Biobehav Rev. 2023 Aug;151:105209. doi: 10.1016/j.neubiorev.2023.105209. Epub 2023 May 5. PMID 37149075
- [Background] Wang Q, Yang Q, Liu X. The microbiota-gut-brain axis and neurodevelopmental disorders. Protein Cell. 2023 Oct 25;14(10):762-775. doi: 10.1093/procel/pwad026. PMID 37166201
- [Background] Tengeler AC, Dam SA, Wiesmann M, Naaijen J, van Bodegom M, Belzer C, Dederen PJ, Verweij V, Franke B, Kozicz T, Arias Vasquez A, Kiliaan AJ. Gut microbiota from persons with attention-deficit/hyperactivity disorder affects the brain in mice. Microbiome. 2020 Apr 1;8(1):44. doi: 10.1186/s40168-020-00816-x. PMID 32238191
- [Background] Elhossiny RM, Elshahawy HH, Mohamed HM, Abdelmageed RI. Assessment of probiotic strain Lactobacillus acidophilus LB supplementation as adjunctive management of attention-deficit hyperactivity disorder in children and adolescents: a randomized controlled clinical trial. BMC Psychiatry. 2023 Nov 9;23(1):823. doi: 10.1186/s12888-023-05324-4. PMID 37946220
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Background] Nanjing consensus on methodology of washed microbiota transplantation. Chin Med J (Engl). 2020 Oct 5;133(19):2330-2332. doi: 10.1097/CM9.0000000000000954. No abstract available. PMID 32701590
- [Background] Bussing R, Fernandez M, Harwood M, Wei Hou, Garvan CW, Eyberg SM, Swanson JM. Parent and teacher SNAP-IV ratings of attention deficit hyperactivity disorder symptoms: psychometric properties and normative ratings from a school district sample. Assessment. 2008 Sep;15(3):317-28. doi: 10.1177/1073191107313888. Epub 2008 Feb 29. PMID 18310593
- [Background] Goyette CH, Conners CK, Ulrich RF. Normative data on revised Conners Parent and Teacher Rating Scales. J Abnorm Child Psychol. 1978 Jun;6(2):221-36. doi: 10.1007/BF00919127. PMID 670589
- [Background] Bruni O, Ottaviano S, Guidetti V, Romoli M, Innocenzi M, Cortesi F, Giannotti F. The Sleep Disturbance Scale for Children (SDSC). Construction and validation of an instrument to evaluate sleep disturbances in childhood and adolescence. J Sleep Res. 1996 Dec;5(4):251-61. doi: 10.1111/j.1365-2869.1996.00251.x. PMID 9065877
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Hooi SL, Dwiyanto J, Rasiti H, Toh KY, Wong RKM, Lee JWJ. A case report of improvement on ADHD symptoms after fecal microbiota transplantation with gut microbiome profiling pre- and post-procedure. Curr Med Res Opin. 2022 Nov;38(11):1977-1982. doi: 10.1080/03007995.2022.2129232. Epub 2022 Oct 7. PMID 36164761